CLINICAL TRIAL: NCT06805695
Title: Long-term Follow-up (LTFU) Study of Participants in Any iECURE Protocol Using an Investigational Product (IP)
Status: Recruiting | Type: Observational
Sponsor: iECURE, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECUR-LTFU
Record Dates: First submitted 2024-12-20; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Ornithine Transcarbamylase Deficiency; Ornithine Transcarbamylase Deficiency Disease; Urea Cycle Disorders, Inborn
Keywords: Amino Acid Metabolism, Inborn Errors; Ammonia; Brain Diseases; Brain Diseases, Metabolic; Brain Diseases, Metabolic, Inborn; Central Nervous System Diseases; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; High Ammonia; Hyperammonemia; Inborn; Inborn Errors; Liver Disease; Liver Transplant; Metabolism; Metabolic Diseases; Metabolism, Inborn Errors; Neonatal; Nervous System Diseases; NH4; Ornithine; Ornithine Transcarbamylase Deficiency; OTC; OTC Deficiency; OTCD; Transcarbamylase; UCD; Urea Cycle Disorders; Long Term Follow Up; Long-Term Follow-Up; LTFU
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease; Urea Cycle Disorders, Inborn; Amino Acid Metabolism, Inborn Errors; Brain Diseases; Brain Diseases, Metabolic; Brain Diseases, Metabolic, Inborn; Central Nervous System Diseases; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Hyperammonemia; Liver Diseases; Metabolic Diseases; Metabolism, Inborn Errors; Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enrolled and Dosed: Previously dosed in a previous iECURE study.
  Interventions: Other: No Intervention
- Enrolled but Not Dosed: Enrolled in a previous iECURE study, but not dosed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
This LTFU is being conducted to assess long-term safety and durability of response in participants dosed with IP in a parent protocol, and to collect longitudinal natural history in enrolled but not dosed participants who also participated in a parent protocol.

DETAILED DESCRIPTION:
This is a 14.5 year LTFU protocol to assess long term safety and clinical response to IP as well as to capture natural disease history of participants not dosed with IP in a parent protocol. No IP is provided as part of this protocol. Participants will remain on standard of care medication as indicated and prescribed by their physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in an iECURE parent protocol and have either completed or discontinued that protocol
2. Participant parent(s)/LAR is willing and able to adhere to the protocol requirements.
3. Consent was obtained by the participants parent(s)/LAR (and participant assent, where applicable), prior to any study-related data being collected.

Exclusion Criteria:

1. Participants who enroll into an interventional drug or gene therapy clinical trial utilizing an IP other than the IP provided in the parent protocol will be excluded from this protocol.

Ages: 7 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All participants from an iECURE parent treatment protocol, whether they received IP or not, will be consented to enter this LTFU study. Enrollment into the LTFU will begin upon either premature discontinuation from, or completion of, the parent treatment protocol.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2041-07 (Estimated); Study Completion 2041-07 (Estimated)

PRIMARY OUTCOMES:
AE and SAE (incidence, severity, seriousness, and relatedness) | Over 14.5 years post dosing with ECUR-506
  Safety
Change from baseline over 14.5 years post infusion in length | Over 14.5 years post dosing with ECUR-506
  Length measured in cenitmeters
Change from baseline over 14.5 years post infusion in weight | Over 14.5 years post dosing with ECUR-506
  Weight measured in kilograms
Urinalysis (Dip Stick) Evaluations | Over 14.5 years post dosing with ECUR-506
  Urinalysis (Dip Stick) will be evaluated to monitor pathological changes to the participants urine and to monitor levels of Specific Gravity, pH, Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen, Nitrite, Leukocyte esterase, red blood cell count, and white blood cell count as they relate to established local lab normal ranges.

SECONDARY OUTCOMES:
qPCR measurement to evaluate the clearance of both vectors in blood over time. | Over 14.5 years post dosing with ECUR-506
  Pharmacokinetics
qPCR measurement to evaluate the clearance of both vectors in saliva over time. | Over 14.5 years post dosing with ECUR-506
  Pharmacokinetics
qPCR measurement to evaluate the clearance of both vectors in urine over time. | Over 14.5 years post dosing with ECUR-506
  Pharmacokinetics
qPCR measurement to evaluate the clearance of both vectors in feces over time. | Over 14.5 years post dosing with ECUR-506
  Pharmacokinetics
Percent Liver Transduction | Over 14.5 years post dosing with ECUR-506
  Pharmacokinetics
Number of hyperammonemic crises (HAC) | Over 14.5 years post dosing with ECUR-506
  Pharmacodynamics and Efficacy
Among participants who experience HAC with associated neurological status change and are hospitalized: Asses daily ammonia levels for duration of hospitalization for each event | Over 14.5 years post dosing with ECUR-506
  Pharmacodynamics and Safety
Among participants who experience HAC with associated neurological status change and are hospitalized: Assess duration of hospitalization for each event. | Over 14.5 years post dosing with ECUR-506
  Pharmacodynamics and Safety
Among participants who experience HAC with associated neurological status change and are hospitalized: Assess requirement for ICU care. | Over 14.5 years post dosing with ECUR-506
  Pharmacodynamics and Safety
Number of HAC with the following severities: a. Mild: adjustment of dietary protein intake and oral scavenger medication b. Moderate: cessation of dietary protein intake and initiation of IV scavenger therapy c. Severe: requirement for hemodialysis | Over 14.5 years post dosing with ECUR-506
  Pharmacodynamics and Safety
Scavenger drug dose per body surface area (BSA) | Over 14.5 years post dosing with ECUR-506
  Efficacy
Protein allowance g/kg | Over 14.5 years post dosing with ECUR-506
  Efficacy
Concentration of blood urea nitrogen measurements | Over 14.5 years post dosing with ECUR-506
  Pharmacodynamics
Time to liver transplant from Day 1 (Parent Protocol) for participants who are dosed and Day -1 (Parent Protocol) for participants who are not dosed to end of study EOS (LTFU Protocol) | Over 14.5 years post dosing with ECUR-506
  Efficacy
Transplant free survival | Over 14.5 years post dosing with ECUR-506
  Efficacy
Time to liver transplant or any cause of death from dosing to EOS. | Over 14.5 years post dosing with ECUR-506
  Efficacy
Overall Survival: Survival measured from Day 1 (Parent Protocol) for participants who are dosed and Day -1 (Parent Protocol) for participants who are not dosed to end of study EOS (LTFU Protocol). | Over 14.5 years post dosing with ECUR-506
  Efficacy
Time to any-cause death from dosing to EOS. Survival measured from Day 1 (Parent Protocol) for participants who are dosed and Day -1 (Parent Protocol) for participants who are not dosed to end of study EOS (LTFU Protocol). | Over 14.5 years post dosing with ECUR-506
  Efficacy

OTHER OUTCOMES:
Number of participants with antibodies to hOTC in blood. | Over 14.5 years post dosing with ECUR-506
  Pharmacodynamics
Number of participants with antibodies to M2PCSK9 in blood. | Over 14.5 years post dosing with ECUR-506
  Pharmacodynamics
Number of participants with antibodies to AAVrh79 in blood. | Over 14.5 years post dosing with ECUR-506
  Pharmacodynamics
Concentration of plasma ammonia | Over 14.5 years post dosing with ECUR-506
  Pharmacodynamics
Concentration of plasma citrulline | Over 14.5 years post dosing with ECUR-506
  Pharmacodynamics
Concentration of plasma glutamine | Over 14.5 years post dosing with ECUR-506
  Pharmacodynamics
Urinary excretion of phenylacetate metabolites. | Over 14.5 years post dosing with ECUR-506
  Urinary phenylactate (mcg/mL), urinary phenylactylglutamine (mcg/mL), urinary phenylacetate/ phenylglutamine ratio.
Urinary excretion of orotic acid metabolites | Over 14.5 years post dosing with ECUR-506
  Urinary orotic acid (mmol/mol creatinine), urinary uracil (mmol/mol creatinine)
Future DNA analysis of WBCs collected in a parent trial may be performed only in the event of an observed genomic safety signal | Over 14.5 years post dosing with ECUR-506
  Safety
Developmental assessments as measured by age-appropriate Bayley Scale of Infant Development IV (BSID-IV) | Over 14.5 years post dosing with ECUR-506
  Total Raw Scores, Growth Score Values (GSVs), and Age Equivalent Scores will be analyzed; Raw Scores range 0-162; GSVs range 428-599; Age Equivalent Scores range 1-42 months; a higher score reflects a higher level of skill.
Kaufman Assessment Battery for Children - Second Edition Normative Update (KABC-II NU) | Over 14.5 years post dosing with ECUR-506
  Total Raw Scores, Growth Score Values (GSVs), and Age Equivalent Scores will be analyzed; Raw Scores range 0-162; GSVs range 428-599; Age Equivalent Scores range 1-42 months; a higher score reflects a higher level of skill.
Quality of life as measured by an age-appropriate Pediatric Quality of Life Inventory Infant Scales | Over 14.5 years post dosing with ECUR-506
  Quality of Life Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: George Diaz, M.D., Ph.D, Study Director — iECURE, Inc.
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided